CLINICAL TRIAL: NCT00760825
Title: An Open Label Post Licensure Trial to Evaluate the Safety and Immunogenicity of Indigenously Manufactured Killed Bivalent (O1 and O139) Whole Cell Oral Cholera Vaccine(Shanchol™)
Brief Title: A Study to Evaluate Safety and Immunogenicity of the Bivalent Killed Whole Cell Oral Cholera Vaccine in Adults and Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Shantha Biotechnics Limited (Industry); Christian Medical College, Vellore, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CH-WC-02
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Vibrio Cholerae
Keywords: cholera; vibrios; oral cholera vaccine
MeSH Terms: conditions — Cholera | interventions — shanchol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental): killed bivalent (O1 and O139)whole cell oral cholera vaccine(Shanchol™)
  Interventions: Biological: killed bivalent (O1 and O139)whole cell oral cholera vaccine

INTERVENTIONS:
Biological: killed bivalent (O1 and O139)whole cell oral cholera vaccine — 1.5 ml given twice orally, 14 days apart
  Other Names: Shanchol™

SUMMARY:
The purpose of this study is to determine whether the killed bivalent (O1 and O139)whole cell oral cholera vaccine(Shanchol™) is safe and effective in the treatment of Vibrio cholerae.

DETAILED DESCRIPTION:
Provision of safe water and food, establishment of adequate sanitation, and implementation of personal and community hygiene constitute the main public health interventions against cholera. These measures cannot be implemented fully in the near future in most cholera-endemic areas. Improvements to water and sanitation require substantial long-term investments, commitment from the local government, and often take years to implement. In the meantime, a safe, effective and affordable vaccine would be a useful tool for cholera prevention and control.

Considerable progress has been made during the last decade in the development of new generation oral vaccines against cholera. These have already been licensed in some countries and are now being considered for wider public health application. Cholera immunization is now recommended for travelers to high risk areas, refugee camps and for outbreak response. Furthermore, expanded use of cholera vaccines may be recommended for endemic areas, where there is increasing demand from both low- and middle-income populations.

Starting in the mid-1980s, following technology transfer from Prof Jan Holmgren, Vietnamese scientists at the National Institute of Hygiene and Epidemiology (NIHE) in Hanoi developed and produced an oral, killed cholera vaccine for the country's public health programs. A two-dose regimen of a first generation monovalent (anti-O1) cholera vaccine produced at US$ 0.10 per dose underwent a field trial in Hue, Vietnam. The study was not formally randomized: the vaccine was assigned on the basis of a systematic allocation scheme and the control group did not receive a placebo. The calculated efficacy against El Tor cholera was 66% in fully immunized adults and children. Protection against non-cholera was assessed and none was found suggesting a non-biased study design. Subsequently, killed 0139 whole cells were added to the Vietnamese vaccine due to the emergence of the new form of epidemic cholera caused by this serogroup. A study found the bivalent vaccine to be safe and immunogenic in adults and children one year and older.

The Vietnamese vaccine has several distinct advantages over the Swedish vaccine. The Vietnamese vaccine confers protection against the El Tor biotype in younger children. And the price of US $0.10 per dose is feasible for public health programs in developing countries, while the Swedish vaccine is prohibitively expensive. Finally, it can be administered without a buffer, while the Swedish vaccine requires a buffer and stricter cold chain requirements.

Since licensure of the oral cholera vaccine in Vietnam, more than 9 million doses have been administered without any report of serious adverse events. The vaccine is produced according to recommended guidelines at the Company for Vaccine and Biological Production No. 1 (VABIOTECH) in Hanoi. VABIOTECH is working towards WHO Good Manufacturing Practices (GMP) certification, which they hope to receive in the next few years. At the same time, the IVI and VABIOTECH have been working to internationalize the Vietnamese vaccine for global use. In order to comply with WHO requirements, the vaccine was reformulated.

Phase II trials of this reformulated killed oral cholera vaccine were performed in SonLa, Vietnam and Kolkata, India where the vaccine was found to be safe and no serious adverse reaction was associated with the vaccine. The vaccine elicited significant vibriocidal antibody responses among vaccinees. In SonLa, 90% of adult recipients seroconverted to V. cholerae O1 following receipt of two doses of the vaccine. In Kolkata, 53% of adults and 80% of children aged 1-17 years developed 4-fold and greater rises in vibriocidal antibodies to V. cholerae O1. Data from Vietnam and India suggest that greater magnitudes in the vibriocidal responses following 2 doses of the vaccine are elicited compared to previous formulations. It has been suggested that this response may correlate with the higher lipopolysaccharide content of the vaccine, a result of changes in its standardization.

A phase III trial of this vaccine is currently underway in Wards 29, 30, and 33 of Kolkata, India. Since this trial is still ongoing, data regarding adverse events still has not been analyzed. As yet no serious adverse reaction has been directly attributed to the vaccine. Surveillance continues in these areas to determine the efficacy of the vaccine.

Through an agreement negotiated by the IVI, VABIOTECH produced the bulk reformulated bivalent vaccine under quality conditions supervised by the IVI. Shantha Biotechnics of India filled and finished the bulk, and obtained regulatory clearance for use of the vaccine in Phase II and III trials in India. In return, the technology for future production of the oral killed bivalent cholera vaccine was transferred to Shantha Biotechnics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged 18-40 years and children aged 1 -17 years who the investigator believes will comply with the requirements of the protocol (i.e. available for follow-up visits and specimen collection).
2. For females of reproductive age, they must not be pregnant (as determined by verbal screening).
3. Written informed consent obtained from the subjects or their parents/guardians, and written assent for children aged 12 - 17 years.
4. Healthy subjects as determined by: Medical history, Physical examination, Clinical judgment of the investigator

Exclusion Criteria:

1. Ongoing serious chronic disease
2. Immunocompromising condition or therapy
3. Diarrhea (3 or more loose/more watery stools within a 24-hour period) 6 weeks prior to enrollment
4. One or two episodes of diarrhea lasting for more than 2 weeks in the past 6 months
5. One or two episodes of abdominal pain lasting for more than 2 weeks in the past 6 months
6. Intake of any anti-diarrhea medicine in the past week
7. Abdominal pain or cramps, loss of appetite, nausea, general ill-feeling or vomiting in the past 24 hours
8. Acute disease one week prior to enrollment, with or without fever. Temperature ≥38ºC (oral) or axillary temperature ≥ 37.5ºC warrants deferral of the vaccination pending recovery of the subject
9. Receipt of antibiotics in past 14 days
10. Receipt of live or killed enteric vaccine in past 4 weeks
11. Receipt of killed oral cholera vaccine

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with diarrhea | 28 days
Proportion of subjects exhibiting 4-fold or greater rises in titers of serum vibriocidal antibodies relative to baseline | 14 days after each dose

SECONDARY OUTCOMES:
Geometric mean serum vibriocidal titers | baseline and 14 days after each dose
Proportion of subjects with any of the following adverse events: immediate reactions, serious adverse events, reactogenicity: headache, vomiting, nausea, abdominal pain/cramps, gas, diarrhea, fever, loss of appetite, general ill feeling | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Venkata R Mohan, M.D., MPH, Principal Investigator — Christian Medical College, Vellore, India
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India

REFERENCES:
- [Derived] Raghava Mohan V, Raj S, Dhingra MS, Aloysia D'Cor N, Singh AP, Saluja T, Kim DR, Midde VJ, Kim Y, Vemula S, Narla SK, Sah B, Ali M. Safety and immunogenicity of a killed bivalent (O1 and O139) whole-cell oral cholera vaccine in adults and children in Vellore, South India. PLoS One. 2019 Jun 18;14(6):e0218033. doi: 10.1371/journal.pone.0218033. eCollection 2019. PMID 31211792